CLINICAL TRIAL: NCT03732105
Title: Randomized Study of Adjuvant Radiotherapy After Curative Resection of Hepatocellular Carcinoma With Narrow Margin (≤1 cm)
Brief Title: Randomized Study of Adjuvant Radiotherapy After Curative Resection of HCC With Narrow Margin (RAISE)
Acronym: RAISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou Medical University (Other); Southern Medical University, China (Other); Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Ming Kuang, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018175
Record Dates: First submitted 2018-11-04; First posted 2018-11-06 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma; Radiotherapy; Hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery-radiotherapy (Experimental): Patients in the surgery-radiotherapy group will receive Intensity Modulated Radiation Therapy (IMRT) at a dose of 50Gy/25fraction after surgery. After radiotherapy, patients will be actively monitored.
  Interventions: Radiation: Surgery-radiotherapy
- Surgery group (No Intervention): Patients in the surgery group will be actively monitored after randomization.

INTERVENTIONS:
Radiation: Surgery-radiotherapy — Patients in the surgery-radiotherapy group will receive Intensity Modulated Radiation Therapy (IMRT) at a dose of 50Gy/25fraction after randomization.
  Arms: Surgery-radiotherapy

SUMMARY:
RAISE is a multicenter randomized controlled trial to assess the efficacy of adjuvant radiotherapy for controlling postsurgical recurrence in HCC patients with narrow margin (≤ 1 cm) after curative resection.

DETAILED DESCRIPTION:
RAISE trial will recruit 148 patients, and they will be randomized (1:1) to two groups (the surgery group and the surgery-radiotherapy group). Random assignment was stratified by the condition of MVI and tumor size. All patients in the surgery-radiotherapy group received Intensity Modulated Radiation Therapy (IMRT) within 1-3 months after surgical resection. The prescription dose was planned at 50 gray in 25 fractions over 5-6 weeks. The trial is to verify whether adjuvant radiotherapy prolongs recurrence-free survival in patients with a narrow resection margin.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 75 years.
2. HCC who underwent R0 resection with pathological confirmation.
3. The narrowest margin is less than or equal to 1 cm.
4. No residual tumors after surgery based on postoperative CT or MR images in 4-6 weeks.
5. ECOG PS ≤ 1.
6. Child-Pugh score 5-7.
7. Expected life expectancy ≥ 6 months.
8. Blood, liver, and kidney functions meet the following criteria: 1)Neutrophil counts ≥ 1.5×109/L; 2)Platelet counts ≥ 60×109/L; 3)Hemoglobin concentration ≥ 90g/L; 4)Serum albumin concentration ≥ 30g/L; 5)Bilirubin ≤ 1.5 × upper limit of normal; 6)AST and ALT < 3× ULN; 7)Extended prothrombin time not exceeding 3s of ULN; 8)Creatinine < 1.5× ULN.

Exclusion Criteria:

1. Preoperative imaging revealed tumor thrombus in the portal vein, hepatic vein, bile duct, or extrahepatic metastasis.
2. The number of tumors ≥4.
3. Pregnant or lactating women or subjects scheduled for contraceptive procedures within 2 years.
4. Patients with concomitant HIV or syphilis infection.
5. Patients with concurrent or other malignancies within 5 years before enrollment.
6. Patients receiving allogeneic organ transplantation.
7. Patients with severe dysfunction of the heart, kidneys or other organs.
8. Participated in clinical trials of other drugs within 12 months before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2018-08-08 (Actual); Primary Completion 2025-08-11 (Estimated); Study Completion 2025-08-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival,RFS | two years
  Defined as the time from randomization until disease recurrence or death from any cause, whichever happens first.

SECONDARY OUTCOMES:
Overall Survival, OS | two years
  Defined as the time from randomization until death from any cause.
Time To Recurrence, TTR | two years
  Defined as the time from randomization until disease recurrence.
Incidence of Treatment-Emergent Adverse Events during the treatment period using Common Terminology Criteria for Adverse Events (CTCAE) (version 4). | two years
  Incidence of Treatment-Emergent Adverse Events during the treatment period using Common Terminology Criteria for Adverse Events (CTCAE) (version 4)causality of Adverse Events (AEs) during the treatment period using Common Terminology Criteria for Adverse Events (CTCAE) (version 4).
health related quality of life | two years
  The quality of life is accessed by EORTC QLQ-C30 (version 3).

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Rodriguez-Peralvarez M, Luong TV, Andreana L, Meyer T, Dhillon AP, Burroughs AK. A systematic review of microvascular invasion in hepatocellular carcinoma: diagnostic and prognostic variability. Ann Surg Oncol. 2013 Jan;20(1):325-39. doi: 10.1245/s10434-012-2513-1. Epub 2012 Nov 13. PMID 23149850
- [Result] Wang WH, Wang Z, Wu JX, Zhang T, Rong WQ, Wang LM, Jin J, Wang SL, Song YW, Liu YP, Ren H, Fang H, Wang WQ, Liu XF, Yu ZH, Li YX. Survival benefit with IMRT following narrow-margin hepatectomy in patients with hepatocellular carcinoma close to major vessels. Liver Int. 2015 Dec;35(12):2603-10. doi: 10.1111/liv.12857. Epub 2015 Jun 3. PMID 25939444
- [Result] Yu W, Wang W, Rong W, Wang L, Xu Q, Wu F, Liu L, Wu J. Adjuvant radiotherapy in centrally located hepatocellular carcinomas after hepatectomy with narrow margin (<1 cm): a prospective randomized study. J Am Coll Surg. 2014 Mar;218(3):381-92. doi: 10.1016/j.jamcollsurg.2013.11.030. Epub 2013 Dec 2. PMID 24559953